CLINICAL TRIAL: NCT01485926
Title: A Phase II Neo-adjuvant Study Assessing TCH (Docetaxel, Carboplatin and Trastuzumab) and TCHL (Docetaxel, Carboplatin, Trastuzumab and Lapatinib) in HER-2 Positive Breast Cancer Patients.
Acronym: TCHL Phase II
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Trials Ireland (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTRIAL-IE (ICORG) 10-05
Record Dates: First submitted 2011-12-02; First posted 2011-12-06 (Estimated); Last update posted 2018-08-06 (Actual); Status verified 2018-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel; Carboplatin; Trastuzumab; Lapatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Docetaxel, Carboplatin and Trastuzumab (Experimental): Arm A- 6 cycles q3weekly Docetaxel (75mg/m²) + Carboplatin (AUC 6) + Trastuzumab 8 mg/kg on day 1 (loading dose) and 6mg/kg for subsequent cycles, q3weekly thereafter. Patients will be scheduled for surgery and will continue to receive Trastuzumab post-operatively 6 mg/kg for one year from 1st dose of Trastuzumab.
  Interventions: Drug: Docetaxel, Carboplatin and Trastuzumab
- Docetaxel, Carboplatin, Trastuzumab and Lapatinib (Experimental): Arm B - 6 cycles q3weekly Docetaxel (75mg/m²) + Carboplatin (AUC 6) + Trastuzumab (8 mg/kg on day 1 (loading dose) and 6mg/kg for subsequent cycles, q3weekly thereafter.) + Lapatinib (1000mg daily) until 1 week prior to surgery. Patients will be scheduled for surgery and will continue to receive Trastuzumab post-operatively 6 mg/kg for one year from 1st dose of Trastuzumab.
  Interventions: Drug: Docetaxel, Carboplatin, Trastuzumab and Lapatinib

INTERVENTIONS:
Drug: Docetaxel, Carboplatin and Trastuzumab — 6 cycles q3weekly Docetaxel (75mg/m²) + Carboplatin (AUC 6) + Trastuzumab 8 mg/kg on day 1 (loading dose) and 6mg/kg for subsequent cycles, q3weekly thereafter. Patients will be scheduled for surgery and will continue to receive Trastuzumab post-operatively 6 mg/kg for one year from 1st dose of Trastuzumab.
  Arms: Docetaxel, Carboplatin and Trastuzumab
Drug: Docetaxel, Carboplatin, Trastuzumab and Lapatinib — 6 cycles q3weekly Docetaxel (75mg/m²) + Carboplatin (AUC 6) + Trastuzumab (8 mg/kg on day 1 (loading dose) and 6mg/kg for subsequent cycles, q3weekly thereafter.) + Lapatinib (1000mg daily) until 1 week prior to surgery. Patients will be scheduled for surgery and will continue to receive Trastuzumab post-operatively 6 mg/kg for one year from 1st dose of Trastuzumab.
  Arms: Docetaxel, Carboplatin, Trastuzumab and Lapatinib

SUMMARY:
The primary objective:

-To assess the efficacy of TCH and TCHL in neo-adjuvant treatment of HER-2 positive breast cancer, using pathological complete response (pCR) as the primary endpoint (Phase II).

Secondary objectives:

* To assess the clinical response rate and overall response rate for docetaxel and carboplatin with trastuzumab alone or trastuzumab combined with lapatinib in HER-2 positive breast cancer.
* To assess the relationship between drug exposure and adverse events.
* To examine potential molecular and pharmacological markers of response to trastuzumab and lapatinib
* To assess Disease-free Survival (DFS) and Overall Survival (OS)
* To determine if prophylactic Loperamide significantly reduces the number of diarrhoea -related adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained prior to any study-related procedures
2. Age > 18 years
3. Histologically proven breast cancer, for which neo-adjuvant chemotherapy and trastuzumab is considered a valid therapeutic strategy.
4. Patients with the following TNM stages (refer to AJCC 7th Edition - Appendix M) of breast cancer are eligible:

   * T2, T3, T4a, T4b, T4c, T4d which is node negative or node positive (histologically or cytologically confirmed) or
   * Any T with lymph node positive disease (histologically or cytologically confirmed)
   * Patients with multifocal tumours are not excluded; T stage assignment must be based on the largest tumour.
   * Patients presenting with bilateral breast cancer are not eligible
5. Tumour HER2/neu positive (3+ by IHC or fluorescence in situ hybridization (FISH) positive)
6. Oestrogen and progesterone receptor status known prior to study entry
7. ECOG performance status score < or equal to 1
8. Cardiac ejection fraction ≥ 50% as measured by echocardiogram or MUGA scan within 3 months prior to randomisation. Note that baseline and on treatment scans should be performed using the same modality and preferably at the same institution
9. The effects of lapatinib on the developing human foetus at the recommended therapeutic dose are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (non-hormonal or barrier method of birth control, abstinence or a vasectomy partner) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

   -If applicable, post-menopausal status will be defined as patients who are amenorrheic for > 1 year or for a shorter duration if FSH, LH and/or oestradiol levels are within the post-menopausal range
10. Patient is accessible and willing to comply with treatment, tissue acquisition and follow up.
11. Formalin-fixed paraffin-embedded tissue available from diagnostic biopsy and/or definitive surgical intervention

    -Where possible fresh frozen tissue will be sought as outlined per protocol.
12. Adequate bone marrow function within 14 days prior to randomisation as defined by the following laboratory values

    1. Absolute neutrophil count ≥ 1.0 x 10^9/L
    2. Haemoglobin ≥ 9.0 g/dL
    3. Platelet count ≥ 100 x 10^9/L
13. Adequate renal function within 14 days prior to randomisation as defined by:

    1. Serum creatinine < or equal to 1.25 x upper limit of normal (ULN), defined by institution
    2. Serum creatinine clearance of > 60 mg/ml/min
14. Adequate hepatic function within 14 days prior to randomisation as defined by:

    1. Total bilirubin < or equal to 1.0 x upper limit of normal (ULN). Patients with Gilbert's syndrome prior to study entry must have total bilirubin <3X ULN.
    2. Alkaline phosphatase and AST/ALT within parameters specified by protocol.
15. Able to swallow and retain oral medication
16. Patients must be deemed potentially operable following neo-adjuvant treatment.

Exclusion Criteria:

1. Prior therapy with systemic cytotoxic chemotherapy Lapatinib or Trastuzumab.
2. Prior taxanes
3. Radiotherapy (Except for radiotherapy localised to radiotherapy to a primary squamous or basal cell skin cancer).
4. Patients with metastatic disease (M1).
5. Concurrent therapy with any other non-protocol anti-cancer therapy
6. History of any other malignancy within the past 5 years, with the exception of non-melanoma skin cancer, in situ carcinoma of the breast (ductal or lobular) or carcinoma-in-situ of the cervix.
7. Current therapy with any hormonal agent such as raloxifene, tamoxifen, or other selective oestrogen receptor modulators (SERMs), either for osteoporosis or prevention of breast cancer. Patients must have discontinued these agents 14 days prior to enrolment.
8. Concurrent treatment with ovarian hormonal replacement therapy. Prior treatment must be stopped prior to enrolment.
9. Pre-existing motor or sensory neurotoxicity of a severity ≥ Grade 2 by NCI-CTCAE version 4.0.
10. Poorly controlled hypertension (e.g. systolic >180mm Hg or diastolic >100mm Hg.)
11. Any history of myocardial infarction, angina pectoris or congestive heart failure. Patients on current therapy for arrythmias are excluded. For other patients with a history of self-limiting cardiac dieases (e.g. pericarditis, temporary secondary arrythmias) more than 1 year must have past prior to enrolment on the study
12. Inflammatory bowel disease or other bowel condition causing chronic diarrhoea, requiring active therapy.
13. Active, uncontrolled infection requiring parenteral antimicrobials or any condition requiring maintenance therapeutic (i.e. non-replacement) doses of corticosteroids.
14. The presence of any other medical or psychiatric disorder that, in the opinion of the treating physician, would contraindicate the use of the drugs in this protocol or place the patient at undue risk for treatment complications
15. Male patients.
16. Patients with known hypersensitivity to Chinese hamster ovary products or other recombinant human or humanized antibodies and/or known hypersensitivity to any of the study drugs or their ingredients (eg, polysorbate 80 in docetaxel)
17. Pregnant women are excluded from this study because lapatinib is member of the 4-anilinoquinazoline class of kinase inhibitors with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with lapatinib, breastfeeding should be discontinued if the mother is treated with lapatinib
18. HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions with lapatinib. Appropriate studies will be undertaken in patients receiving combination anti-retroviral therapy when indicated.
19. Patients with GI tract disease resulting in an inability to take oral medication, malabsorption syndrome, a requirement for IV alimentation, prior surgical procedures affecting absorption, uncontrolled inflammatory GI disease (e.g., Crohn's, ulcerative colitis).
20. Concomitant requirement for medication classified as CYP3A4 inducers or inhibitors as defined in Table 2.
21. Have current active hepatic or biliary disease (with exception of patients with Gilbert's syndrome, asymptomatic gallstones, liver metastases or stable chronic liver disease per investigator assessment)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2010-10; Primary Completion 2014-09 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
pathological complete response | 5 months

CONTACTS AND LOCATIONS:
Locations (11):
- Ireland (11):
  - St James's Hospital, Dublin, Leinster
  - St Vincent's University Hospital, Dublin, Leinster
  - Bon Secours Hospital, Cork
  - Cork University Hospital, Cork
  - Beaumont Hospital, Dublin
  - Mater Misericordiae University and Private Hospitals, Dublin
  - Galway University Hospital, Galway
  - Letterkenny General Hospital, Letterkenny
  - Mid-Western Regional Hospital, Limerick
  - Sligo General Hospital, Sligo
  - Waterford Regional Hospital, Waterford

REFERENCES:
- [Derived] Crown J, Eustace AJ, Collins DM, Keane M, Coate L, Kennedy J, O'Reilly S, Kelly C, O'Connor M, Martin M, Murphy C, Duffy K, Walshe J, Gullo G, Mahgoub T, Alvarez-Iglesias A, Parker I, Donachie V, Teiserskiene A, Madden SF, Moulton B, O'Donovan N, Hennessy BT. TCHL - a phase II neo-adjuvant study assessing TCH (docetaxel, carboplatin and trastuzumab) and TCHL (docetaxel, carboplatin, trastuzumab and lapatinib) in HER-2 positive breast cancer patients: a 5-year follow-up with serum biomarker analysis. Acta Oncol. 2025 Jun 5;64:751-760. doi: 10.2340/1651-226X.2025.43143. PMID 40468999
- [Derived] Gaynor N, Blanco A, Madden SF, Moran B, Fletcher JM, Kaukonen D, Ramirez JS, Eustace AJ, McDermott MSJ, Canonici A, Toomey S, Teiserskiene A, Hennessy BT, O'Donovan N, Crown J, Collins DM. Alterations in immune cell phenotype and cytotoxic capacity in HER2+ breast cancer patients receiving HER2-targeted neo-adjuvant therapy. Br J Cancer. 2023 Oct;129(6):1022-1031. doi: 10.1038/s41416-023-02375-y. Epub 2023 Jul 28. PMID 37507543
- [Derived] Toomey S, Eustace AJ, Fay J, Sheehan KM, Carr A, Milewska M, Madden SF, Teiserskiene A, Kay EW, O'Donovan N, Gallagher W, Grogan L, Breathnach O, Walshe J, Kelly C, Moulton B, Kennedy MJ, Gullo G, Hill AD, Power C, Duke D, Hambly N, Crown J, Hennessy BT. Impact of somatic PI3K pathway and ERBB family mutations on pathological complete response (pCR) in HER2-positive breast cancer patients who received neoadjuvant HER2-targeted therapies. Breast Cancer Res. 2017 Jul 27;19(1):87. doi: 10.1186/s13058-017-0883-9. PMID 28750640